CLINICAL TRIAL: NCT03297580
Title: Itch and Clinacal Caracteristics in Systemic Sclerosis
Acronym: SCLERODERMIE
Status: Completed | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: SCLERODERMIE
Record Dates: First submitted 2017-09-20; First posted 2017-09-29 (Actual); Last update posted 2017-09-29 (Actual); Status verified 2017-09

CONDITIONS: Pruritus; Systemic Sclerosis
MeSH Terms: conditions — Pruritus; Scleroderma, Systemic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Systemic sclerosis (SSc) has heterogeneous symptoms and significant medical morbidity. Recently, itch was described as a symptom of SSc (prevalence of 42,6%). To the investigators knowledge, no study yet has examined the clinical features of itch neither had used a specific itch-related quality of life (QoL) scales in patients with SSc. The objectives were to evaluate the prevalence of pruritus, its characteristics and its impact on the QoL in those patients.

In this descriptive study, patients followed for SSc in the departments of dermatology, rheumatology, internal medicine and pulmonology at the University Hospital of Brest were included. Participants received a questionnaire including questions about the clinical features of pruritus and 2 scores (5-D itch scale, ItchyQol).

ELIGIBILITY:
Inclusion Criteria:

* aged more than 18 years
* followed for systemic sclerosis since 2000, in the departments of dermatology, rheumatology, internal médicine or pneumology at the University Hospital of Brest.

Exclusion Criteria:

* lower than 18 years
* refusal to participate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with a systemic sclerosis followed in the University Hospital of Brest
Sampling Method: Non-Probability Sample
Enrollment: 61 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-03-31 (Actual); Study Completion 2016-03-31 (Actual)

PRIMARY OUTCOMES:
Pruritus | Day 1 (questionnaire sent to patient)
  Pruritus: yes/no

SECONDARY OUTCOMES:
Characteristics of the systemic sclerosis | Day 1 (questionnaire sent to patient)
  Duration of the disease
Brest questionnaire | Day 1 (questionnaire sent to patient)
  questions about the chronology, location, intensity, disruption of daily activities, characteristics of scratching and other associated sensations
5-D itch scale | Day 1 (questionnaire sent to patient)
  Validated questionnaire about severity of pruritus using five items (duration, intensity, evolution, impact on daily activities, localisation)
ItchyQol scale | Day 1 (questionnaire sent to patient)
  questionnaire about quality of life linked to pruritus
Characteristics of the systemic sclerosis | Day 1 (questionnaire sent to patient)
  treatments,
Characteristics of the systemic sclerosis | Day 1 (questionnaire sent to patient)
  topography of skin involvement (limited or diffuse systemic sclerosis)

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU de Brest, Brest, France